CLINICAL TRIAL: NCT04918277
Title: Ultrasound Assessment of Gastric Volume and Aspiration Risk Evaluation in the Fasted Pediatric Cerebral Palsy Patients
Brief Title: Gastric Volume in the Fasted Pediatric Cerebral Palsy Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, JiWon Han, assistant professor, Seoul National University Bundang Hospital
Other Study IDs: L-2021-365
Record Dates: First submitted 2021-06-03; First posted 2021-06-08 (Actual); Last update posted 2021-06-08 (Actual); Status verified 2021-06

CONDITIONS: Aspiration, Respiratory; Cerebral Palsy
MeSH Terms: conditions — Respiratory Aspiration; Cerebral Palsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Assessment of gastric volume — Measuring the cross-sectional area of stomach in supine and right lateral decubitus

SUMMARY:
In children with cerebral palsy, the gastric volume is measured through ultrasound after fasting before surgery to evaluate whether the risk of aspiration is higher than that of the general population.

ELIGIBILITY:
Inclusion Criteria:

* Patients with cerebral palsy under the age of 18 undergoing surgery under general anesthesia

Exclusion Criteria:

* Levin tube or gastrostomy tube in situ
* Decline to participate

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients with cerebral palsy under the age of 18 undergoing surgery under general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 38 (Estimated)
Dates: Start 2021-06-05 (Estimated); Primary Completion 2022-05-30 (Estimated); Study Completion 2022-08-30 (Estimated)

PRIMARY OUTCOMES:
gastric volume | preoperative 1 days to postoperative 1 days
  Volume = -7.8 + (3.5 x RLD CSA) + 0.127 X age (months)

SECONDARY OUTCOMES:
Grade of gastric fullness | preoperative 1 days to postoperative 1 days
  Grade 0: Neither in supine, right lateral decubitus / Grade 1: stomach content only in lateral decubitus , Grade 2: Both in supine, lateral decubitus

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Spencer AO, Walker AM, Yeung AK, Lardner DR, Yee K, Mulvey JM, Perlas A. Ultrasound assessment of gastric volume in the fasted pediatric patient undergoing upper gastrointestinal endoscopy: development of a predictive model using endoscopically suctioned volumes. Paediatr Anaesth. 2015 Mar;25(3):301-8. doi: 10.1111/pan.12581. Epub 2014 Dec 11. PMID 25495405